CLINICAL TRIAL: NCT07217795
Title: Developing a Telehealth Intervention for Alcohol and Trauma Among LGBTQ+ People
Brief Title: Recovery Through Inhibitory Learning, Self-Efficacy Building, Problem Solving, and Community Building
Acronym: RISE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rhode Island (Other)
Collaborators: Rhode Island Foundation (Other)
Responsible Party: Principal Investigator, Jillian Scheer, Assistant Professor, University of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2310793
Record Dates: First submitted 2025-08-12; First posted 2025-10-16 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Alcohol Use Disorder (AUD); PTSD
Keywords: LGBTQ; cognitive behavioral therapy; expressive writing; PTSD; alcohol use; telehealth
MeSH Terms: conditions — Alcoholism; Stress Disorders, Post-Traumatic; Alcohol Drinking

STUDY DESIGN:
Intervention Model Description: The overall objective of this project is to adapt and pilot test a remotely delivered alcohol-focused cognitive behavioral therapy (CBT) intervention and trauma-focused expressive writing (EW) intervention addressing social determinants of unhealthy alcohol use and traumatic stress among sexual minority women (SMW; e.g., lesbian, bisexual) and transgender and gender-diverse (TGD) people. The Recovery through Inhibitory Learning, Self-Efficacy Building, Problem-Solving, and Community Building (RISE) intervention will integrate adapted CBT modules on assertiveness, problem-solving in high-risk situations, and connecting with others-shown to reduce unhealthy alcohol use-with a brief EW intervention tailored to SMW and TGD people. The four specific Unified Protocol (CBT) modules that will be adapted for the current study are 1) Psychoeducation, goal setting, motivational enhancement; 2) Mindful emotional awareness; 3) Cognitive flexibility; and 4) Countering emotional-driven behaviors.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RISE (Experimental): Description: Participants receive the RISE intervention, a remotely delivered CBT + Expressive Writing program.
  Intervention: Behavioral: RISE (CBT + Expressive Writing)
  Interventions: Behavioral: CBT + expressive writing
- Control: Wait-List Control (Other): Participants are placed on a wait-list and offered the RISE intervention after the study period.
  Interventions: Behavioral: Wait-List Control

INTERVENTIONS:
Behavioral: CBT + expressive writing — This study will test a remotely delivered intervention combining Cognitive Behavioral Therapy (CBT) and Expressive Writing (EW) to address unhealthy alcohol use and traumatic stress among sexual minority women (SMW; e.g., lesbian, bisexual women) and transgender and gender-diverse (TGD) individuals. The intervention, called Recovery through Inhibitory Learning, Self-Efficacy Building, Problem-Solving, and Community Building (RISE), integrates CBT modules on assertiveness, problem-solving in high-risk situations, and building social connections with a brief EW program tailored to SMW and TGD participants. Four modules from the Unified Protocol (UP), a transdiagnostic CBT approach, will be adapted: (1) psychoeducation, goal setting, and motivational enhancement; (2) mindful emotional awareness; (3) cognitive flexibility; and (4) countering emotion-driven behaviors.
  Arms: RISE
Behavioral: Wait-List Control — Participants assigned to the wait-list will not receive active treatment during the study period but will be offered the RISE intervention afterward.
  Arms: Control: Wait-List Control

SUMMARY:
This is a two-part study to develop and test a brief, virtual therapy program for lesbian, gay, bisexual, transgender, and queer (LGBTQ+) people who have experienced trauma and use alcohol.

Phase 1: You'll be invited to share your perspective to help make the program relevant, inclusive, and affirming.

Phase 2: You may have the opportunity to try the adapted program by receiving free virtual therapy with LGBTQ+-affirming therapists.

ELIGIBILITY:
Aim 1: Sexual Minority Women and Transgender and Gender Diverse Individuals -Not meeting inclusion criteria

Aim 1: Providers

-Not meeting inclusion criteria

Aim 2: Sexual Minority Women and Transgender and Gender Diverse Individuals

* Not meeting inclusion criteria OR any of the following:
* Reporting current mental health treatment ≥1 day/month
* Receiving Cognitive Behavioral Therapy (CBT) in the past 3 months (note: participants are not ineligible if they seek concomitant care after enrollment)
* Reporting current alcohol or drug use disorder treatment, except mutual self-help (e.g., Alcoholics Anonymous) or current PTSD/trauma-focused treatment
* Need for alcohol detoxification, defined as score ≥15 on the adapted self-report Clinical Institute Withdrawal Assessment for Alcohol - Revised (CIWA-Ar)
* Active psychosis, defined as score ≥1 on the psychosis subscale of the Behavior and Symptom Identification Scale - Revised (BASIS-R)
* Active mania, defined as score ≥6 on the Altman Self-Rating Mania Scale (ASRM)
* Active suicidality, defined as score ≥22 on the Suicidal Ideation Attributes Scale (SIDAS)
* Currently legally mandated to attend treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-11-30 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Posttraumatic Stress Disorder Diagnosis and Severity using the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) | Baseline: Past 30 days 1-week Follow-up: Past 1 week
  Posttraumatic Stress Disorder (PTSD) will be assessed using the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5), a clinician-administered interview that evaluates Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) PTSD criteria. It provides both a total severity score (0-80) and a dichotomous diagnosis (present/absent).
  Units of Measure: Total score (0-80); diagnosis status (yes/no)
Posttraumatic Stress Disorder Symptom Severity using the PTSD Checklist for DSM-5 (PCL-5) | Baseline: Past 30 days 1-week Follow-up: Past 1 week
  Posttraumatic Stress Disorder (PTSD) symptom severity will be assessed using the PTSD Checklist for DSM-5 (PCL-5), a 20-item self-report measure. Items are rated on a 5-point Likert scale from 0 ("Not at all") to 4 ("Extremely"), with a total score range of 0-80; higher scores indicate greater PTSD symptom severity. A score of 33 or higher suggests probable PTSD. Units of Measure: Total score (0-80).
Hazardous drinking levels | Baseline: Past 3 months 1-week Follow-up: Past 1 week
  Structured Clinical Interview for DSM-5 - Substance Use Disorders Module (SCID-5-SUD)
  Description: Structured Clinical Interview for DSM-5 - Substance Use Disorders Module (SCID-5-SUD) will be used to assess the presence and severity of substance use disorders (SUDs). The SCID-5-SUD is a semi-structured clinical interview administered by trained personnel to determine whether a participant meets Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) diagnostic criteria for a substance use disorder (e.g., alcohol, cannabis, opioids, stimulants). For each substance, the SCID-5-SUD evaluates 11 diagnostic criteria, including impaired control, social impairment, risky use, and pharmacological indicators. Severity is categorized based on the number of criteria endorsed: mild (2-3), moderate (4-5), or severe (6 or more).
  Units of Measure: Dichotomous diagnosis status (yes/no); severity level (mild, moderate, severe) if applicable
Change in average weekly drinking quantity | Baseline: Past 30 days 1-week Follow-up: Past 1 week
  The Timeline Followback (TLFB) method will be used to assess daily alcohol consumption over the past 30 days. Participants report the number of standard drinks consumed each day, using a calendar-assisted structured interview format. Data are used to calculate total number of drinking days, total drinks consumed, average drinks per drinking day, and number of heavy drinking days (4+ drinks for women, 5+ for men). This measure provides a reliable estimate of recent alcohol use patterns and is widely used in clinical and research settings.
  Units of Measure: Number of drinking days, total drinks, drinks per drinking day,
Change in heavy drinking frequency | Baseline: Past 30 days 1-week Follow-up: Past 1 week
  Description: Alcohol use will be assessed using a six-item self-report measure evaluating past-week drinking frequency, quantity, and risky use. Items include: frequency of drinking (scored 0-6), maximum number of drinks in 24 hours (scored 1-10), typical number of drinks per drinking day (scored 1-10), total number of drinks per week (scored 1-11), and frequency of binge drinking (defined as 4 or more drinks in one occasion) and high-intensity drinking (defined as 8 or more drinks in one occasion), both scored 0-6.
  In addition, the Timeline Followback (TLFB) method will be used to assess daily alcohol use over the past 30 days. The TLFB captures number of drinking days, total number of drinks, average drinks per drinking day, and number of heavy drinking days.
  Units of Measure: Item scores range 0-6, 1-10, or 1-11; TLFB outcomes include days and number of drinks.

SECONDARY OUTCOMES:
Depression symptoms | Baseline: Past 1 week 1-week Follow-up: Past 1 week
  Title: Depression Severity and Impairment (ODSIS)
  Description:
  The Overall Depression Severity and Impairment Scale (ODSIS) is a 5-item self-report measure assessing the frequency and intensity of depressive symptoms, as well as related distress and functional impairment. Each item is rated on a 0-4 scale, with total scores ranging from 0 to 20. Higher scores indicate greater severity of depression and impairment. The ODSIS is sensitive to clinical change and has strong psychometric properties.
  Units of Measure: Total score (0-20)
Anxiety symptoms | Baseline: Past 1 week 1-week Follow-up: Past 1 week
  Title: Anxiety Severity and Impairment (OASIS) Description: The Overall Anxiety Severity and Impairment Scale (OASIS) is a 5-item self-report measure assessing the frequency and intensity of anxiety symptoms, as well as related avoidance, distress, and functional impairment. Each item is rated on a 0-4 scale, with total scores ranging from 0 to 20. Higher scores indicate greater anxiety severity and impairment. The OASIS is brief, transdiagnostic, and sensitive to treatment-related change.
  Units of Measure: Total score (0-20)
Perceived Stress | Baseline: Past 30 days 1-week Follow-up: Past 1 week
  Title: Perceived Stress (PSS-10)
  Description: The Perceived Stress Scale-10 (PSS-10) is a 10-item self-report measure that assesses the degree to which individuals perceive their life situations as stressful over the past month. Each item is rated on a 0-4 scale, with total scores ranging from 0 to 40. Higher scores indicate greater perceived stress. The PSS-10 is widely used and has demonstrated strong reliability and validity across populations.
  Units of Measure: Total score (0-40)
Suicidality | Baseline: Past 30 days 1-week Follow-up: Past 1 week
  Title: Suicidal Ideation Attributes Scale (SIDAS) Description: The Suicidal Ideation Attributes Scale (SIDAS) is a 5-item self-report measure assessing the severity of suicidal thoughts over the past 30 days, including frequency, controllability, closeness to attempt, associated distress, and functional interference. Each item is rated on a 0-10 scale, with total scores ranging from 0 to 50. Higher scores indicate more severe suicidal ideation. A score of 21 or above indicates high risk and warrants clinical attention.
  Units of Measure: Total score (0-50)
Readiness to change | Baseline: At baseline assessment 1-week Follow-up: At 1-week follow-up assessment
  Title: Readiness to Change Alcohol Use (Readiness Ruler)
  Description: The Readiness Ruler is a single-item self-report measure assessing how ready a person feels to change their alcohol use. Participants rate their readiness on a scale from 0 ("not at all ready") to 10 ("completely ready"). Higher scores indicate greater motivation to change drinking behavior. This tool is commonly used in brief interventions and motivational interviewing.
  Units of Measure: Score (0-10)
Change in maximum number of drinks on any day | Baseline: Past 30 days 1-week Follow-up: Past 1 week
  Title: Maximum Drinks in a 24-Hour Period (Past Week) Description: This single-item self-report measure assesses the maximum number of alcoholic drinks consumed within a 24-hour period during the past week. Participants select one of 10 ordinal response options ranging from 1 ("1 drink") to 10 ("36 drinks or more"). Higher scores reflect greater peak alcohol consumption.
  Units of Measure: Score (1-10)
Alcohol-related consequences | Baseline: Past 90 days 1-week Follow-up: Past 1 week
  Title: Alcohol-Related Consequences (Short Inventory of Problems-2R)
  Description: The Short Inventory of Problems-2R (SIP-2R) is a 15-item self-report measure assessing adverse consequences of alcohol use across five domains: physical, interpersonal, intrapersonal, impulse control, and social responsibility. Items are rated based on how often each consequence occurred in the past 3 months using a 4-point scale from 0 ("never") to 3 ("daily or almost daily"). Total scores range from 0 to 45, with higher scores indicating greater alcohol-related problems.
  Units of Measure: Total score (0-45)
Alcohol craving | Baseline: Past 1 week 1-week Follow-up: Past 1 week
  Title: Alcohol-Related Consequences (Short Inventory of Problems-2R)
  Description: The Short Inventory of Problems-2R (SIP-2R) is a 15-item self-report questionnaire measuring negative consequences of alcohol use over the past 3 months across five domains: physical, interpersonal, intrapersonal, impulse control, and social responsibility. Each item is rated on a 4-point scale from 0 ("never") to 3 ("daily or almost daily"). Total scores range from 0 to 45, with higher scores indicating more frequent or severe alcohol-related problems.
  Units of Measure: Total score (0-45)
Alexithymia | Baseline: At baseline assessment 1-week Follow-up: At 1-week follow-up assessment
  Title: Alexithymia Severity (Perth Alexithymia Questionnaire)
  Description: Alexithymia will be assessed using the 24-item Perth Alexithymia Questionnaire (PAQ), a self-report measure evaluating difficulties identifying and describing feelings across positive and negative emotions. The focus will be on the negative-difficulty identifying feelings and negative-difficulty describing feelings subscales. Items are rated on a 7-point Likert scale from 1 ("Strongly disagree") to 7 ("Strongly agree"). Higher scores indicate greater alexithymia. Total and subscale scores will be calculated by summing relevant items.
  Units of Measure: Total and subscale scores (higher scores indicate greater alexithymia)
Anxiety sensitivity | Baseline: At baseline assessment 1-week Follow-up: At 1-week follow-up assessment
  Title: Anxiety Sensitivity (SSASI)
  Description: Anxiety sensitivity will be assessed using the Short Scale Anxiety Sensitivity Index (SSASI), a 5-item self-report measure evaluating concerns about the physical, cognitive, and social consequences of anxiety-related sensations. Items include fears of bodily sensations, cognitive control, and social evaluation (e.g., "When I tremble in the presence of others, I fear what people might think of me"). Each item is rated on a 5-point scale from 0 ("very little") to 4 ("very much"). Total scores are calculated by summing all items, with higher scores indicating greater anxiety sensitivity.
  Units of Measure: Total score (0-20)
Negative emotionality | Baseline: At baseline assessment 1-week Follow-up: At 1-week follow-up assessment
  Title: Negative Emotionality Big Five Inventory-2 (BFI-2)
  Description: Negative emotionality will be assessed using the Big Five Inventory-2 (BFI-2) self-report form. Participants rate 12 items describing emotional tendencies (e.g., mood swings, worry, sadness) on a 5-point scale from 1 ("disagree strongly") to 5 ("agree strongly"). Reverse-scored items (r) are included to assess emotional stability. Subscale and total negative emotionality scores are calculated as the mean of relevant items, with higher scores indicating greater negative emotionality.
  Units of Measure: Mean score (1-5)
Posttraumatic maladaptive beliefs scale | Baseline: At baseline assessment 1-week Follow-up: At 1-week follow-up assessment
  Title: Posttraumatic Maladaptive Beliefs (PMBS)
  Description: Posttraumatic beliefs will be assessed using the Posttraumatic Maladaptive Beliefs Scale (PMBS), a self-report measure evaluating negative cognitions and beliefs following trauma. Items assess domains such as self-blame, mistrust of others, and perceptions of threat or vulnerability. Participants rate each item on a Likert scale (e.g., 1 = "strongly disagree" to 5 = "strongly agree"), with higher scores indicating more maladaptive posttraumatic beliefs. Total and subscale scores can be calculated to assess the severity and domain-specific patterns of trauma-related cognitions.
  Units of Measure: Total and subscale scores (higher scores indicate greater maladaptive beliefs)
Dissociation | Baseline: Past 1-week 1-week Follow-up: Past 1-week
  Title: Dissociative Experiences Brief Dissociative Experiences Scale-B (DES-B Modified)
  Description: Dissociative experiences will be assessed using the 8-item Modified Brief Dissociative Experiences Scale (DES-B). Participants rate each item based on experiences over the past 7 days, using a 5-point scale: 0 = "Not at all," 1 = "Once or twice," 2 = "Almost every day," 3 = "About once a day," and 4 = "More than once a day." Total scores range from 0 to 32, with higher scores indicating greater severity. An average total score is calculated by dividing the total score by 8, yielding a 0-4 scale corresponding to none, mild, moderate, severe, or extreme dissociation.
  Units of Measure: Total score (0-32) and average score (0-4)
Brief experiential avoidance questionarraire | Baseline: At baseline assessment 1-week Follow-up: At 1-week follow-up assessment
  Title: Experiential Avoidance Brief Experiential Avoidance Questionnaire (BEAQ)
  Description: Experiential avoidance will be assessed using the Brief Experiential Avoidance Questionnaire (BEAQ), a self-report measure evaluating the tendency to avoid or escape unwanted internal experiences. Participants rate items on a 6-point scale from 1 ("strongly disagree") to 6 ("strongly agree"). Item 6 is reverse-scored, and total scores are calculated by summing all items, with higher scores indicating greater experiential avoidance.
  Units of Measure: Total score (sum of items; higher scores indicate greater avoidance)
Coping | Baseline: At baseline assessment 1-week Follow-up: At 1-week follow-up assessment
  Title: Coping Strategies (Brief Coping Orientation to Problems Experienced [COPE])
  Description: Coping strategies will be assessed using the Brief Coping Orientation to Problems Experienced (COPE), a 28-item self-report measure evaluating how individuals respond to stressors over the past 30 days. Items are rated on a 4-point scale: 1 = "I haven't been doing this at all," 2 = "I've been doing this a little bit," 3 = "I've been doing this a medium amount," and 4 = "I've been doing this a lot." Subscale scores are calculated as the mean of two items per subscale, including indicators of avoidance coping (self-distraction, denial, behavioral disengagement) and other coping strategies. Higher scores indicate greater use of the specific coping strategy.
  Units of Measure: Mean subscale scores (1-4)
Emotion regulation | Baseline: At baseline assessment 1-week Follow-up: At 1-week follow-up assessment
  Title: Emotion Regulation Difficulties Short Form (Difficulties in Emotion Regulation Scale Short Form [DERS-SF])
  Description: Emotion regulation difficulties will be assessed using the Difficulties in Emotion Regulation Scale Short Form (DERS-SF), an 18-item self-report measure evaluating challenges in managing emotions, including nonacceptance of emotional responses and difficulties engaging in goal-directed behavior. Items are rated on a 5-point scale from 1 ("almost never") to 5 ("almost always"), with the acceptance items reverse-scored. Mean scores are calculated, with higher scores indicating greater difficulties in emotion regulation.
  Units of Measure: Mean score (1-5)
Self-Compassion | Baseline: At baseline assessment 1-week Follow-up: At 1-week follow-up assessment
  Title: Self-Compassion Scale (SCS - Self-Kindness, Common Humanity, Mindfulness Subscales)
  Description: Self-compassion will be assessed using the Self-Compassion Scale (SCS), focusing on the self-kindness, common humanity, and mindfulness subscales. Participants rate items on a 5-point scale from 1 ("almost never") to 5 ("almost always"), indicating how often they engage in the behaviors described. Mean scores are calculated for each subscale, with higher scores reflecting greater self-compassion.
  Units of Measure: Mean score (1-5)
Loneliness | Baseline: At baseline assessment 1-week Follow-up: At 1-week follow-up assessment
  Title: Loneliness (University of California, Los Angeles [UCLA] Loneliness Scale - Short Form)
  Description: Loneliness will be assessed using the 3-item short form of the UCLA Loneliness Scale. Participants indicate how often they experience feelings of lacking companionship, feeling left out, or feeling isolated from others. Items are rated on a 4-point Likert scale: 1 = "Never," 2 = "Rarely," 3 = "Sometimes," and 4 = "Often."
  Units of Measure: Total score (range: 3-12), with higher scores indicating greater loneliness.
Social support | Baseline: At baseline assessment 1-week Follow-up: At 1-week follow-up assessment
  Title: Perceived Social Support (Multidimensional Scale of Perceived Social Support [MSPSS])
  Description: Perceived social support will be assessed using the Multidimensional Scale of Perceived Social Support (MSPSS), a 12-item self-report measure evaluating support from family, friends, and a significant other. Items are rated on a 7-point scale from 1 ("Very Strongly Disagree") to 7 ("Very Strongly Agree"). Total scores are calculated by summing all items, with higher scores indicating greater perceived social support. Subscale scores can also be calculated for each support source.
  Units of Measure: Total score (12-84) and subscale scores
LGBTQ+ Community connection | Baseline: At baseline assessment 1-week Follow-up: At 1-week follow-up assessment
  Title: LGBTQ+ Community Connection (Lesbian, Gay, Bisexual Positive Identity Measure [LGB-PIM])
  Description: Connection to the LGBTQ+ community will be assessed using the 5-item LGBTQ+ Community Connection subscale of the Lesbian, Gay, Bisexual Positive Identity Measure (LGB-PIM). Items assess feelings of support, visibility, inclusion, connection, and positive networking within the LGBTQ+ community. Participants rate each item on a 7-point scale from 1 ("Strongly Disagree") to 7 ("Strongly Agree"). Mean scores are calculated, with higher scores indicating stronger perceived connection to the LGBTQ+ community.
  Units of Measure: Mean score (1-7)
Positive and Negative Affect | Baseline: Past 4 weeks 1-week Follow-up: Past 1 week
  Title: Positive and Negative Affect (PANAS)
  Description: Mood will be assessed using the 10-item Positive and Negative Affect Schedule (PANAS), past-week version. Participants rate the extent to which they have experienced various positive and negative emotions (e.g., distressed, nervous, irritable) over the past 7 days. Items are rated on a 5-point scale, with higher mean scores indicating greater levels of positive or negative affect. Separate mean scores are calculated for the positive affect and negative affect scales.
  Units of Measure: Mean score (1-5) for positive affect and negative affect
Physical health | Baseline: Past 2 weeks 1-week Follow-up: Past 1 week
  Title: Physical Health (World Health Organization Quality of Life-BREF [WHOQOL-BREF])
  Description: Physical health will be assessed using the World Health Organization Quality of Life-BREF (WHOQOL-BREF) physical health item. Participants rate the extent to which physical pain has interfered with their ability to perform daily activities over the past week. Items are rated on a 5-point scale: 1 = "Not at all," 2 = "A little," 3 = "A moderate amount," 4 = "Very much," 5 = "An extreme amount." Negatively framed items are reverse-scored, and total or summed scores reflect better physical health when higher.
  Units of Measure: Summed score (1-5 per item)
LGBTQ-Hypervigilance | Baseline: Past 12 months 1-week Follow-up: Past 1 week
  Title: LGBTQ+ Hypervigilance
  Description: Hypervigilance related to LGBTQ+ identity will be assessed using the LGBTQ-Hypervigilance Scale, a self-report measure evaluating heightened alertness or vigilance in public or social settings. Participants rate each item based on experiences in the past week on a 7-point scale from 1 ("Strongly Disagree") to 7 ("Strongly Agree"), with higher scores indicating greater hypervigilance.
  Units of Measure: Total score or mean item score (higher scores indicate greater LGBTQ+ hypervigilance)
Lesbian, Gay, Bisexual Identity Scale | Baseline: At baseline assessment 1-week Follow-up: At 1-week follow-up assessment
  Title: Sexual Minority Identity (Lesbian, Gay, Bisexual Identity Scale - Internalized Homonegativity & Concealment Motivation)
  Description: Sexual minority identity will be assessed using the Lesbian, Gay, and Bisexual Identity Scale (LGBIS), focusing on the Internalized Homonegativity (IH) and Concealment Motivation (CM) subscales. Participants rate items on a 6-point scale from 1 ("Disagree strongly") to 6 ("Agree strongly") reflecting their current experiences as a sexual minority. Subscale scores are calculated by averaging relevant items, with higher scores indicating greater internalized homonegativity or stronger motivation to conceal one's sexual orientation.
  Units of Measure: Mean subscale scores (1-6)
Cannabis use | Baseline: Past 3 months 1-week Follow-up: Past 1 week
  Title: Cannabis Use (Cannabis Use Disorder Identification Test - Revised [CUDIT-R])
  Description:
  Cannabis use over the past week will be assessed using a single item from the Cannabis Use Disorder Identification Test - Revised (CUDIT-R). Participants indicate whether they have used cannabis in the past 7 days. Responses are coded as 1 = "Yes" and 0 = "No."
  Units of Measure: Binary (Yes = 1, No = 0)
Other drug use | Baseline: Past 1 month 1-week Follow-up: Past 1 week
  Title: Past-Week Substance Use (National Survey on Drug Use and Health [NSDUH])
  Description: Past-week substance use will be assessed using items adapted from the 2020 National Survey on Drug Use and Health (NSDUH). Participants report: (1) the number of days they smoked cigarettes in the past 7 days (0-30), and (2) the average number of cigarettes smoked per day on those days (coded 1-7: less than 1, 1, 2-5, 6-15, 16-25, 26-35, more than 35). Participants also report the number of days they used other illicit drugs or misused prescription drugs in the past week (0-30 days). Higher values indicate greater substance use.
  Units of Measure: Number of days (0-30) for each substance; average cigarettes per day (1-7)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rhode Island, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No
Data from this study will not be shared due to the sensitive nature of the information collected and the pilot status of the project. Additionally, data sharing is not required by the study's funder.